CLINICAL TRIAL: NCT02787291
Title: A Clinical Evaluation of the Durata or Optisure High Voltage Leads and Ellipse VR ICD Undergoing Magnetic Resonance Imaging, an Investigational Device Exemption (IDE) Study
Brief Title: A Clinical Evaluation of the Durata or Optisure High Voltage Leads and Ellipse VR ICD Undergoing MRI, an IDE Study
Acronym: MRI Ready IDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-CRD768
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Implantable Defibrillator User

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ellipse VR ICD and Durata/Optisure lead (Other): Pts with Ellipse VR ICD and Durata or Optisure RV lead implanted for at least 60 days will receive a non-diagnostic MRI scan of head and chest region
  Interventions: Device: Ellipse VR ICD and Durata/Optisure lead

INTERVENTIONS:
Device: Ellipse VR ICD and Durata/Optisure lead — Non-diagnostic MRI Scan sequence of head and chest

SUMMARY:
To demonstrate safety and efficacy of the Durata or Optisure high voltage lead and Ellipse VR ICD in an MRI environment.

DETAILED DESCRIPTION:
The intent of this IDE study is to evaluate the safety and efficacy of the Durata or Optisure lead and Ellipse VR ICD that have undergone an MRI scan. The patient population under study includes patients indicated for or who have been implanted with a Durata or Optisure lead and an Ellipse VR ICD.

ELIGIBILITY:
Inclusion Criteria:

* Are implanted with the Durata or Optisure lead for at least 60 days (can include patients with Durata or Optisure lead for > 60 days OR patients with a new Ellipse VR ICD and/or Durata/Optisure lead implanted for at least 60 days
* Are implanted with an Ellipse VR ICD pectorally
* Be willing to undergo an elective MRI scan without sedation NOTE: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the patient can communicate with site personnel during the MRI scan
* Capture threshold is stable < 2.5V @ 0.5ms
* Ventricular sensing is measurable (patient has underlying rhythm > 30bpm) and the sensing amplitude is > 4mV
* Be able to provide informed consent for study participation (legal guardian or legally authorized representative is NOT acceptable)
* Be willing and able to comply with the prescribed follow-up tests and procedures
* Are not contraindicated for an MRI scan (per the MRI Screening Form)

Exclusion Criteria:

* Have a competitor's MRI compatible endocardial lead implanted or capped
* Have another existing active implanted medical device, e.g., neurostimulator, infusion pump, etc., that has MR labeling that will not allow the MRI scans per this protocol to be completed.
* Have a lead revision of the Durata/Optisure lead occur < 60 days of the baseline visit
* Have other non-MRI compatible device or material implanted NOTE: MRI compatible knee replacements, hip replacements, stents, etc. may be included as long as the labeling of these devices allow MRI scans conducted per this protocol NOTE: MRI compatible mechanical, prosthetic, and bioprosthetic heart valves may be included as long as the labeling of these devices allow for MRI scans conducted per this protocol NOTE: Non-removable dental implants may be included
* Have a lead extender, adaptor, or capped/abandoned lead
* Enrolled or intend to participate in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug or additional testing beyond standard of care procedures), which could confound the results of this trial as determined by SJM.
* Pregnant or planning to become pregnant during the duration of the subject's participation in the study
* Have a life expectancy of less than 12 months due to any condition
* Patients with exclusion criteria required by local law (e.g., age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saman Nazarian, MD, Study Chair — Johns Hopkins University Hospital
Locations (32):
- United States (26):
  - John C. Lincoln North Mountain Hospital, Phoenix, Arizona
  - Central Cardiology, Bakersfield, California
  - Scripps Health, La Jolla, California
  - Florida Hospital, Orlando, Florida
  - Athens Regional Medical Center, Athens, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Medical Consultants, Muncie, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Providence Hospital, Southfield, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - St. Francis, Roslyn, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Samaritan Heart & Vascular Institute, Corvallis, Oregon
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - West Virginia University Hospital, Morgantown, West Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
  - Cardiac Rhythm Specialists, S.C., Milwaukee, Wisconsin
- Semmelweis University, Budapest, Hungary
- Poland (3):
  - Szpital Kliniczny Premienienia Panskiego, Poznan, Silesian Voivodeship
  - American Heart of Poland SA, Tychy, Silesian Voivodeship
  - Carint Scanmed Sp. z.o.o., Krakow, Voivode
- Hospital Universitario de Salamanca, Salamanca, Castellon, Spain
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nazarian S, Cantillon DJ, Woodard PK, Mela T, Cline AM, Strickberger AS; MRI Ready Investigators. MRI Safety for Patients Implanted With the MRI Ready ICD System: MRI Ready Study Results. JACC Clin Electrophysiol. 2019 Aug;5(8):935-943. doi: 10.1016/j.jacep.2019.05.010. Epub 2019 Jun 26. PMID 31439295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
Started | 227
Completed | 227
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 207
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 201
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 21
  United States | 113
  Poland | 64
  United Kingdom | 11
  Spain | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MRI Scan Related Complications
Description: The primary safety endpoint is the number of participants that had an Ellipse ICD and/or a Durata or Optisure lead complication from the day the MRI scan occurred to the 1-month visit. A complication is defined as a serious adverse device effect that requires an invasive intervention or leads to death.
Time Frame: MRI scan to 1 month post MRI scan
Population: Of 227 subjects enrolled, 209 subjects completed the pre-MRI scan visit. Of the 209 subjects, 4 subjects did not have eligible study leads, 3 withdrew before 1-month post MRI scan visit and 4 missed 1-month post MRI scan visit. Therefore, 198 subjects who completed 1-month post MRI scan were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
Number analyzed (Participants) | 198
Participants | 0

2. Primary Outcome: Percentage of Participants With Ventricular Capture Threshold ≤ to 0.5V
Description: Percentage of participants of Durata or Optisure (RV) leads implanted with the Ellipse VR ICD with capture threshold increase of ≤ 0.5V at 0.5ms from pre-MRI scan to 1 month post-MRI scan.
Time Frame: pre-MRI scan to 1 month post MRI scan
Population: Of 227 subjects enrolled, 209 subjects completed the pre-MRI scan visit. Of the 209 subjects, 4 did not have eligible study leads, 13 were missing capture threshold measurements, 3 withdrew before the 1-month post MRI scan visit and 2 missed the 1-month post MRI scan visit. Therefore, 187 subjects were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
Number analyzed (Participants) | 187
Participants | 0

3. Primary Outcome: Percentage of Participants With Ventricular Sensing Amplitude Decrease of ≤ 50% From Pre-MRI Scan to 1 Month Post MRI Scan
Description: Percentage of Participants with Durata or Optisure RV leads implanted with the Ellipse VR ICD with sensing amplitude decrease of ≤ 50% from pre-MRI scan to 1 month post MRI scan.
Time Frame: pre-MRI scan to 1 month post MRI scan
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
Number analyzed (Participants) | 198
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 month post MRI scan
Description: Protocol defined ADE (Adverse Device Effects), SADEs (Serious Adverse Device Effects), UADE (Unanticipated Adverse Device Effects), and USADEs (Unanticipated Serious Adverse Device Effects) were collected in this trial and were adjudicated by a Clinical Events Committee
Arm/Group | Ellipse VR ICD and Durata/Optisure Lead
All-Cause Mortality (participants affected / at risk) | 2/227
Serious Adverse Events (participants affected / at risk) | 0/227
Other Adverse Events (participants affected / at risk) | 0/227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT02787291/Prot_SAP_ICF_000.pdf